CLINICAL TRIAL: NCT05729061
Title: Analysis of Human Movement With Assistive Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orthocare Innovations, LLC (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: AD-001; R44HD097826 (NIH)
Record Dates: First submitted 2023-01-05; First posted 2023-02-15 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Limb Loss; Limb Weakness; Limb Paralysis; Movement Disorders
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Participant with normal assistive device (No Intervention): Normal assistive device refers to the habitual assistive device that may be prescribed by a provider of care or no assistive device if the individual does not normally use.
- Participant with intervention (Other): Intervention refers to investigational assistive devices or commercially available assistive devices that individuals may use during this study.
  Interventions: Device: Assist-Knee; Device: Prosthetic Knee; Device: Prosthetic Ankle; Device: Prosthetic Foot; Device: Ankle-Foot Orthosis

INTERVENTIONS:
Device: Assist-Knee — Investigational prosthetic knee-ankle device
  Arms: Participant with intervention
Device: Prosthetic Knee — Commercially available prosthetic knee devices
  Arms: Participant with intervention
Device: Prosthetic Ankle — Commercially available prosthetic ankle devices
  Arms: Participant with intervention
Device: Prosthetic Foot — Commercially available prosthetic foot devices
  Arms: Participant with intervention
Device: Ankle-Foot Orthosis — Commercially available ankle-foot orthosis devices
  Arms: Participant with intervention

SUMMARY:
The purpose of this research is to evaluate how people move about in different settings with different assistive devices or components, and to understand how people interact with different assistive technologies. Individuals that have limb weakness, limb paralysis, limb loss, and movement disorders are often provided assistive devices such as prostheses and orthoses to assist with mobility or use assistive technologies for purposes such as to regain muscle strength or retrain movements. It is important to understand the impact of these different assistive technologies on human movement for technology improvement and in preparation for commercialization.

Because this research focuses on evaluating how different people move about in different settings with different assistive devices/components, there are different activities that may take place. These activities have been classified as (1) Movement Analysis in the Laboratory, (2) Movement Analysis Outside the Laboratory, (3) Usability Testing, and (4) Focus Groups. Each participant may or may not complete the same activities as the other participants. Each participant may or may not complete all of the activities. Participants may complete the activities more than once.

ELIGIBILITY:
Inclusion Criteria for Nondisabled Participants:

* Age 18 - 90 years
* Has bilateral normal range of motion
* Able to perform a variety of movement activities
* Able to communicate and write individual perceptions in English
* Able to provide written informed consent
* Participants that will use a treadmill during data collection must also be able to walk independently and safely on a treadmill

Exclusion Criteria for Nondisabled Participants:

* Health issues (e.g., confounding injury, musculoskeletal, or cognitive) or other issues (e.g., transportation or schedule issues) that limit effective participation and/or may not represent a nondisabled condition
* Pregnancy
* Not able to read and understand English

Inclusion Criteria for Participants with a Disability:

* Age 18 - 90 years
* Has a condition or diagnosis that results in limb weakness, limb paralysis, limb loss, or movement disorders
* Medically stable
* Has stable balance
* Able to perform a variety of movement activities
* Able to communicate and write individual perceptions in English
* Able to provide written informed consent
* Participants that will use a treadmill during data collection must also be able to walk independently and safely on a treadmill
* Able to safely complete the movements being tested and/or safely use the assistive devices being tested

Exclusion Criteria for Participants with a Disability:

* Health issues (e.g., confounding injury, musculoskeletal, or cognitive) or other issues (e.g., transportation or schedule issues) that limit effective participation and/or may result in mixed effects of multiple sources of disability
* Pregnancy
* Not able to read and understand English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-11-28 (Estimated); Study Completion 2024-11-28 (Estimated)

PRIMARY OUTCOMES:
Walking Speed with no intervention | Collection at baseline
  Walking speed determined over 8 meters of walking
Walking Speed with intervention | Collection immediately after acclimation with intervention
  Walking speed calculated over 8 meters of walking

SECONDARY OUTCOMES:
Time to Complete Sit-to-Stand with no intervention | Collection at baseline
  The amount of time, measured in seconds, needed by the subject to complete the sit-to-stand transition. At least three trials of the sit-to-stand maneuver are collected for each participant using a motion analysis system. Average and standard deviation of the time to complete the sit-to-stand transition are calculated for each participant. The start of the transition will be determined by participant initiation; the end of the transition will be determined by the participant reaching full knee extension.
Time to Complete Sit-to-Stand with intervention | Collection immediately after acclimation with intervention
  The amount of time, measured in seconds, needed by the subject to complete the sit-to-stand transition. At least three trials of the sit-to-stand maneuver are collected for each participant using a motion analysis system. Average and standard deviation of the time to complete the sit-to-stand transition are calculated for each participant. The start of the transition will be determined by participant initiation; the end of the transition will be determined by the participant reaching full knee extension.
Timed Up and Go (TUG) Test | Collection at baseline
  The Timed Up and Go (TUG) test is a validated timed functional test that involves standing up from a chair, walking forward for 3 meters, turning around, walking back to the chair for 3 meter, and sitting down. Each participant will complete the TUG test for three trials. Time is measured using a stopwatch. Average and standard deviation of the time to complete the TUG test are calculated for each participant.
Timed Up and Go (TUG) Test with intervention | Collected immediately after acclimation with intervention
  The Timed Up and Go (TUG) test is a validated timed functional test that involves standing up from a chair, walking forward for 3 meters, turning around, walking back to the chair for 3 meter, and sitting down. Each participant will complete the TUG test for three trials. Time is measured using a stopwatch. Average and standard deviation of the time to complete the TUG test are calculated for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Arabian, PhD, Principal Investigator — Orthocare Innovations, LLC
Locations (1):
- Orthocare Innovations, LLC, Edmonds, Washington, United States

IPD SHARING:
Plan to Share IPD: No